CLINICAL TRIAL: NCT05640310
Title: Prospective Study to Validate the Clinical Accuracy of Norbert Device to Measure Body Temperature
Status: Withdrawn | Type: Observational
Why Stopped: Internal decision made by Norbert Health
Sponsor: Norbert Health (Industry)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: NCP-0001
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Healthy; Febrile Illness
Keywords: medical device; validation; febrile; thermometer; body temperature; Norbert Device; Norbert Health
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Norbert Device — The Norbert Device (ND) is a contactless, noninvasive device that provides measurements of body temperature, oxygen saturation (SpO2), and pulse rate.

SUMMARY:
The study will evaluate the clinical bias and clinical repeatability of measuring body temperature using the Norbert Device (ND).

DETAILED DESCRIPTION:
The study design is based on the ISO 80601-2-56, Clause 201.102 for adjusted mode clinical thermometers. The study is designed to be a non-randomized, non-blinded single arm design to evaluate the clinical accuracy of the ND's temperature measurement compared to a standard FDA 510(k)-cleared reference clinical thermometer (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 22 years of age
* Ability to provide signed informed consent, and/or have a legally authorized representative (LAR) willing to provide informed consent on behalf of the subject
* ESI score of 3-5

Exclusion Criteria:

* Use of medications known to affect body temperature (for example, antipyretics, barbiturates, thyroid preparations, antipsychotics, etc.) within 3 hours of the study procedure
* Recent immunization within seven days of the study procedure
* Pregnancy
* ESI score of 1-2

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted within an Emergency Department where each subject is assigned an Emergency Severity Index (ESI) score. Only subjects with ESI scores ranging from 3-5 will be recruited for the study to prevent intervening with standard patient care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Bias | Up to 1 hour
  Clinical Bias will be evaluated by comparing the first recorded measurement using ND with the corresponding measurement recorded by the RCT. The bias is calculated per IEC 80601-2-56, Clause 201.103.3.
Limits of Agreement | Up to 1 hour
  Limits of Agreement (LOA) will be calculated using all three measurements by the ND and the corresponding measurements by the RCT. The LOA is calculated per IEC 80601-2-56, Clause 201.103.4.
Clinical Repeatability | Up to 1 hour
  Clinical Repeatability is calculated by a pooled standard deviation of the triplicate measurements over the entire population of subjects. The method to calculate Clinical Repeatability is per IEC 80601-2-56, Clause 201.102.5.

IPD SHARING:
Plan to Share IPD: No